CLINICAL TRIAL: NCT04163562
Title: A Multicenter Double-blind, Randomized, Placebocontrolled Phase I/II Study to Determine the Safety, Tolerability, Potential Efficacy and Dose Finding of INP20, an Oral Formulation for Treatment of Immunotherapy in Peanut-allergic Patients
Brief Title: Oral Immunotherapy for Peanut Allergic Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InnoUp Farma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INP20-01
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INP20 (Oral Immunotherapy) (Experimental)
  Interventions: Drug: INP20
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INP20 — Part A: Oral INP20 administration at ascending doses once daily for 2 weeks. Part B: Two doses of oral INP20 derived from Part A once daily for 6 months.
  Arms: INP20 (Oral Immunotherapy)
Drug: Placebo — Part A: Oral placebo administration onces daily for 2 weeks. Part B: Oral placebo administration onces daily for 6 months.
  Arms: Placebo

SUMMARY:
Multicenter, double-blind, randomized, placebo-controlled phase I/II study to determine the safety, tolerability, potential efficacy and dose finding of INP20, an oral immunotherapy in peanut-allergic patients. The overall study design consists of two sequential periods of Part A and Part B.

Part A is a dose escalation study in patients from 12 to 65 years old with a history of immediate hypersensitive reaction to peanut protein. Six diferent oral-dose of INP20 will be administered to 6 cohorts of patients once daily for 2 weeks.

Part B is a 6-month double-blind, placebo-controlled, randomized and parallel groups study. Patients will be randomized in a 1:1:1 ratio into three (3) different treatment groups, including placebo and the two doses of peanut protein selected from Part A. They will recieve INP20 once daily for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* The presence of specific IgE to peanuts (a positive skin prick test to peanuts (diameter of wheal > 3.0 mm) and a positive peanut IgEs [CAP-FEIA] > 0.35 kUA/L.
* A history of significant clinical symptoms occurring within 60 minutes after ingesting peanuts.
* Have a positive double-blind placebo-controlled food challenge (DBPCFC) to peanut at a cumulative dose of less than 10 grams of peanut protein.
* Provide signed informed consent for the participation in the study.
* Have self-injectable epinephrine available at home and be trained on its proper use.
* Potentially fertile women must agree to be sexually inactive or to use appropriate contraceptive measures for the duration of the study and for 1 month afterward.

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by respiratory distress with cyanosis, hypoxemia (O2 Sat <92%) or, in the absence of other clinical records, severe dyspnea; hypotension with or without loss of consciousness; or relaxation of sphincters.
* Currently participating in another study using an investigational new drug.
* Participation in any interventional study, specific oral or sublingual immunotherapy building up phase for the treatment of food allergy in the past 12 months.
* Allergic to placebo ingredients or reacts to any dose of placebo during study entry DBPCFC.
* Patients allergic to corn food.
* Poor control or persistent activation of severe atopic dermatitis.
* Moderate to severe persistent asthma.
* Prior intubation/mechanical ventilation for asthma.
* Currently being treated with greater than medium daily doses of inhaled corticosteroids (fluticasone >500 μg per day, ciclesonide >400 μg per day or budesonide >800 μg per day) or montelukast.
* Chronic gastrointestinal diseases.
* Primary or secondary immunodeficiency.
* Have a severe reaction at initial DBPCFC (life-threatening anaphylaxis or reaction requiring hospitalization).
* Chronic use of beta blockers, angiotensin converting enzyme inhibitors, or monoamine oxidase inhibitors, proton pump inhibitors, H2-bloquers, prokinetic drugs and laxatives.
* Inability to discontinue antihistamines for 7 days before skin testing and oral food challenges (OFCs).
* Patients diagnosed with other serious food allergies defined as those who have required intubation and/or ICU admission.
* Women of childbearing potential (unless they are using highly effective methods of contraception during dosing and for at least 1 month after stopping medication), who are pregnant, planning to become pregnant, or breastfeeding.
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study may also exclude a participant from the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate, severity, and relationship to treatment of adverse events (AEs) and serious adverse events (SAEs) | Week 4 and Week 25
  Safety of the investigational product
Number of patients experiencing any dose limiting toxicity (DLT) | Week 2
  Tolerability of the investigational product

SECONDARY OUTCOMES:
Change in Immunoglobulin G subtype (IgG4) and basophil activation on the BAT (basophil activation test). | Week 4
  Pharmacodynamics
Differences in reaction thresholds (challenge test) to peanut of treatment groups versus the placebo after 6 months of INP20 treatment. | Week 24
  Efficacy of the investigational product

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ferrer, PhD, MD, Principal Investigator — Clinica Universidad de Navarra; Ana Tabar, PhD, MD, Principal Investigator — Complejo Hospitalario de Navarra
Locations (2):
- Spain (2):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospittalario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Undecided